CLINICAL TRIAL: NCT00507949
Title: Randomized Trial,Comparative With Placebo, Double Blind, to Evaluate the Effect of the Treatment With 320 mg/d of Megestrol Acetate in Patients With Severe Chronic Obstructive Pulmonary Disease (COPD) and Loss of Body Weight. Pilot Study
Brief Title: Study to Evaluate the Effect of Megestrol Acetate in Severe Chronic Obstructive Pulmonary Disease With Loss of Weight
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rottapharm Spain (Industry)
Responsible Party: Anna Anguera, Research Manager, Madaus, S.A.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BO-EC-EPOC-01; EudraCT number:2005-005148-16
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; body weight; megestrol acetate; cytokines
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Body Weight | interventions — Megestrol Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Megestrol acetate: sachets of granulated 160 mg. Dose: 160 mg/b.i.d. Duration 8 weeks
  Interventions: Drug: Megestrol acetate
- 2 (Placebo Comparator): The placebo is the excipient of the experimental drug.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Megestrol acetate — Sachets of 160 mg of granulated. Dosage 160 mg /b.i.d. Duration 8 weeks.
  Arms: 1
Drug: placebo — sachets of granulate of 160 mg. Dosage 160 mg b.i.d. Duration 8 weeks.
  Arms: 2

SUMMARY:
The purpose of this trial is to study the effect of megestrol acetate in the gain of body weight in patients with severe Chronic obstructive pulmonary disease in order to improve the survival of the patients.

DETAILED DESCRIPTION:
It has been demonstrated that the body weight measured as a Body mass index (BMI)is an independent risk factor of mortality in the severe COPD.It seems to be one influence of inflammatory factors in the development of denutrition in these patients.

The use of especial diets has no so good results in the aim to improve the weight, being necessary to complement with muscular rehabilitation or anabolic products. The megestrol acetate has demonstrated good results in a short period of time, nevertheless the studies are scarce.

The beneficial effects of the megestrol acetate seems to be mediated by cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnose of COPD (criteria ATS/ERS 2004)
* Clinical stability more than 3 months
* Smokers or ex-smokers of more than > 10 boxes/year than do not modify their smoking habit during the study.
* FEV1 (post-bronchodilator) < 50%. FEV1/FVC ≤ 70
* Negative answer to bronchodilator(≤ 20% del FEV1 o ≤ 200 ml.after 400 mcg.de salbutamol inhaled)
* BMI < 21 Kg/m2 ó BMI 21-25 Kg/m with loss weight of 5% of the habitual body weight in the last 3 months, without other reason that could explain it independently of the COPD.

Exclusion Criteria:

* Use of nasogastric catheter
* Concomitant treatment with steroid, anabolics or other progestagens.
* Loss of body weight related with other causes: hyperthyroidism, enteral malnutrition ( Crohn disease...), neoplasias,etc
* Treatment with Megestrol Acetate in the last 6 months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-10; Primary Completion 2009-04 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To demonstrate if the Megestrol Acetate administered in dose of 320 mg/d could produce a significative increase of body weight in patients with severe COPD with loss of weight without any known reason in the last 3 months. | 8 weeks

SECONDARY OUTCOMES:
Evaluate if the gain of weight is correlated with an improvement of the functional respiratory parameters | 8 weeks
Evaluate if the gain of weight is related with an improvement in the quality of life of the patients. | 8 weeks
Evaluate the changes in the inflammatory parameters (IL-6, TNF alfa...)and nutritional ones (Albumin and prealbumin) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Herrejon Alberto, MD, Principal Investigator — Hospital Universitario Dr. Peset, Valencia
Locations (1):
- Neumology Service of the Hospital Universitario Dr. Peset, Valencia, Valencia, Spain

REFERENCES:
- [Result] Herrejon A, Palop J, Inchaurraga I, Lopez A, Banuls C, Hernandez A, Blanquer R, Estan N, Anguera A. [Low doses of megestrol acetate increase weight and improve nutrition status in patients with severe chronic obstructive pulmonary disease and weight loss]. Med Clin (Barc). 2011 Jul 23;137(5):193-8. doi: 10.1016/j.medcli.2011.02.016. Epub 2011 Apr 27. Spanish. PMID 21524765